CLINICAL TRIAL: NCT06859489
Title: Active aGeing And Personalised Service's Ecosystem
Brief Title: Active aGeing And Personalised Service's Ecosystem (AGAPE) Aims to Implement an Advanced Technology Platform That Provides Services to the Elderly, Formal and Informal Caregivers, and Caregiving Organizations
Acronym: AGAPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: MEDEA SRL (Unknown); Carol Davila University of Medicine and Pharmacy (Other); Caritas Diocesana de Coimbra (Unknown); Be-Com (Unknown); SenLab d.o.o. (Unknown); Umana Persone (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AGAPE
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Older People; Digital Health Literacy
Keywords: active and healthy ageing; digital health literacy; older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Four categories of end users will be involved:
  1. Primary end users (i.e., older adults);
  2. Secondary end users, in the figure of informal caregivers (i.e., relatives and friends of the elderly);
  3. Secondary end users, in the figure of formal caregivers (i.e., social and health workers with different professional trainings, such as nurses, home care workers, geriatricians etc...);
  4. Tertiary end users (i.e., care organizations, local authorities, municipalities).
  The Agape platform will offer a series of customized and integrated services to meet the needs of end users, including:
  1. promotion of a healthy and active lifestyle;
  2. socialization services;
  3. digital health literacy service.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- primary end-users (Experimental): The Agape platform will offer a series of customized and integrated services to meet the needs of end users, including:
  1. promotion of a healthy and active lifestyle;
  2. socialization services;
  3. digital health literacy service.
  Interventions: Device: Active aGeing And Personalised service's Ecosystem (AGAPE)
- formal caregiver (Other): formal caregivers are social operators with different background. The service provides support to formal caregivers in defining and updating the patient's activity plan over time, ensuring it adapts to their needs.
  Interventions: Device: Active aGeing And Personalised service's Ecosystem (AGAPE)
- informal caregiver (Other): Informal caregivers will be able to receive notifications of any anomalies on their devices and, if necessary, draw the attention of the formal caregiver.
  Interventions: Device: Active aGeing And Personalised service's Ecosystem (AGAPE)
- Tertiary end users (Other): Tertiary end users (i.e., care organizations, local authorities, municipalities).
  The Agape platform will offer a series of customized and integrated services to meet the needs of end users, including:
  1. promotion of a healthy and active lifestyle;
  2. socialization services;
  3. digital health literacy service.
  Interventions: Device: Active aGeing And Personalised service's Ecosystem (AGAPE)

INTERVENTIONS:
Device: Active aGeing And Personalised service's Ecosystem (AGAPE) — The experimental protocol is structured into two phases:
  Phase 1 (pre-pilot) - Preliminary assessment of the functionality and usability of the AGAPE platform by older adults and caregivers, divided into:
  Living lab: Three sessions to progressively explore and test the platform and its services, including workshop activities.
  Testing phase: Use of the platform in the home environment of older adults for one month.
  Phase 2 (pilot study) - Evaluation of the platform's impact on the daily lives of older adults, caregivers, and care organizations, with a 12-month involvement for each user.

SUMMARY:
AGAPE aims to implement an advanced technology platform that provides services to older adults, formal and informal caregivers, and caregiving organizations.

DETAILED DESCRIPTION:
AGAPE aims to promote an active and healthy lifestyle in the over-65 population and, in parallel, to improve the quality of life of caregivers (by reducing the burden of care), while also overcoming the possible digital literacy gap of users. The advantage of the AGAPE platform is to offer users highly personalized services based on their needs and digital capabilities, and innovative technologies integrated with each other that fit within the spatial services already available in local ecosystems. The project involves an impact-by-design approach that engages older people, caregivers, and managers of care organizations in a co-creation strategy. In addition, the solutions offered by the AGAPE platform will be extensively tested in a preliminary pre-validation phase in order to effectively meet the needs of end users.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Ability to understand the rationale and characteristics of the study and to provide informed consent
* Low level of frailty, indicated by a score <5 on the Rockwood Clinical Frailty Scale (Rockwood et al., 2005)
* Absence of moderate to severe cognitive impairment, indicated by a Mini-Mental State Examination (MMSE) score ≥ 24 (adjusted score; Folstein, 1975)
* Absence of severe comorbidities and clinically relevant diseases

Exclusion Criteria:

* Age below 65 years
* Inability to provide informed consent for participation in the study
* High level of frailty (Rockwood Clinical Frailty Scale > 5)
* Presence of cognitive impairment (adjusted MMSE score < 24)
* Diagnosed anxiety and depression
* Presence of severe disability and serious health conditions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | From the enrollment to the end of treatment at 12 months (T2)
  Innovation adoption profile transition of the older adult, innovation adoption profile transition of the caregiver, evaluation of usability and technostress levels of the older adult and their respective caregivers in relation to the AGAPE platform, assessed using the SUS scale and the Technostress questionnaire throughout the different phases of the study.
  Answer: 1 (strongly disagree) - 5 (strongly agree). Minimum= 10 ; Maximum= 50.
System Usability Scale (SUS) | From the enrollment to 6 months (T1)
  Innovation adoption profile transition of the older adult, innovation adoption profile transition of the caregiver, evaluation of usability and technostress levels of the older adult and their respective caregivers in relation to the AGAPE platform, assessed using the SUS scale and the Technostress questionnaire throughout the different phases of the study.
  Answer: 1 (strongly disagree) - 5 (strongly agree). Minimum= 10 ; Maximum= 50.
System Usability Scale (SUS) | From the enrollment to 1 month (T0)
  Innovation adoption profile transition of the older adult, innovation adoption profile transition of the caregiver, evaluation of usability and technostress levels of the older adult and their respective caregivers in relation to the AGAPE platform, assessed using the SUS scale and the Technostress questionnaire throughout the different phases of the study.
  Answer: 1 (strongly disagree) - 5 (strongly agree). Minimum= 10 ; Maximum= 50.
Ad Hoc socio-demographic questionnaire | From the enrollment to 6 months (T1)
  the aim of the questionnaire is recording the socio-demographic charateristics of the sample
Ad Hoc socio-demographic questionnaire | From the enrollment to 12 months (T2)
  the aim of the questionnaire is recording the socio-demographic charateristics of the sample
Ad Hoc socio-demographic questionnaire | From the enrollment to 1 month (T0)
  the aim of the questionnaire is recording the socio-demographic charateristics of the sample
TechnoStress Questionnaire | From the enrollment to 12 months (T2)
  it's a psychological questionnaire designed to measure the level of stress related to the use of technology.
TechnoStress Questionnaire | From the enrollment to1 month (T0)
  it's a psychological questionnaire designed to measure the level of stress related to the use of technology
TechnoStress Questionnaire | From the enrollment to 6 months (T1)
  it's a psychological questionnaire designed to measure the level of stress related to the use of technology
Questionnaire for Innovation Adoption | From the enrollment to1 month (T0)
  it explores how and why individuals decide to embrace or reject innovation such as technology
Questionnaire for Innovation Adoption | From the enrollment to 6 months (T1)
  it explores how and why individuals decide to embrace or reject innovation such as technology
Questionnaire for Innovation Adoption | From the enrollment to 12 months (T2)
  it explores how and why individuals decide to embrace or reject innovation such as technology
EQ-5D-5L | From the enrollment to1 month (T0)
  this questionnaire explores the quality of life for european samples. Answer: 1 (no problems) to 5 (extreme problems).
EQ-5D-5L | From the enrollment to 12 months (T2)
  this questionnaire explores the quality of life for european samples. Answer: 1 (no problems) to 5 (extreme problems).
EQ-5D-5L | From the enrollment to 6 months (T1)
  this questionnaire explores the quality of life for european samples. Answer: 1 (no problems) to 5 (extreme problems).
UCLA Loneliness Scale | From the enrollment to 6 months (T1)
  this scale is used for investigate the loneliness of the sample. Answer: 0 (Never) to 3 (Often).
UCLA Loneliness Scale | From the enrollment to1 month (T0)
  this scale is used for investigate the loneliness of the sample. Answer: 0 (Never) to 3 (Often).
UCLA Loneliness Scale | From the enrollment to 12 months (T2)
  this scale is used for investigate the loneliness of the sample. Answer: 0 (Never) to 3 (Often).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Firenze, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided